CLINICAL TRIAL: NCT01293032
Title: Choosing Neoadjuvant Chemotherapy Versus Hormonal Therapy for Breast Cancer Based on Gene Expression Profile
Brief Title: Hormone Therapy Or Chemotherapy Before Surgery Based on Gene Expression Analysis in Treating Patients With Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MCC-13311; NCI-2010-02342 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); P30CA016059 (NIH)
Record Dates: First submitted 2011-02-07; First posted 2011-02-10 (Estimated); Results first posted 2016-07-12 (Estimated); Last update posted 2016-07-12 (Estimated); Status verified 2016-06

CONDITIONS: Ductal Breast Carcinoma in Situ; Lobular Breast Carcinoma in Situ; Stage II Breast Cancer; Stage IIA Breast Cancer; Stage IIB Breast Cancer; Stage IIIA Breast Cancer; Stage IIIB Breast Cancer
Keywords: Estrogen Receptor Positive; Progesterone Receptor Positive; HER2/Neu Negative; Breast Cancer
MeSH Terms: conditions — Carcinoma, Intraductal, Noninfiltrating; Breast Carcinoma In Situ; Breast Neoplasms | interventions — Neoadjuvant Therapy; Gene Expression Profiling; Tamoxifen; Aromatase Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Group 1 (RS < 11) (Experimental): Patients with a Recurrence Score (RS) less than 11 (RS <11) are assigned to Group 1, neoadjuvant hormonal therapy either tamoxifen (pre-menopausal women) or an aromatase inhibitor (post-menopausal women) for 4-6 months in the absence of disease progression or unacceptable toxicity.
  Treatment:
  * Neoadjuvant therapy
  * Therapeutic conventional surgery
  * Laboratory biomarker analysis/Correlative studies
  * Gene Expression Analysis/ Oncotype DX Gene Expression Profiling System
  * Hormonal therapy:
    * Tamoxifen Citrate (pre-menopausal women) OR
    * Aromatase Inhibition Therapy (post-menopausal women)
  Interventions: Procedure: Neoadjuvant Therapy; Procedure: Therapeutic Conventional Surgery; Other: Laboratory Biomarker Analysis; Genetic: Gene Expression Analysis; Drug: Tamoxifen Citrate; Drug: Aromatase Inhibition Therapy
- Group 2 Arm 1 (RS 11-25) (Experimental): Patients with an intermediate RS (11-25) assigned to Group 2. Randomized to Arm 1, neoadjuvant hormonal therapy as in Group 1.
  Treatment:
  * Neoadjuvant therapy
  * Therapeutic conventional surgery
  * Laboratory biomarker analysis/Correlative studies
  * Gene Expression Analysis/ Oncotype DX Gene Expression Profiling System
  * Hormonal therapy:
    * Tamoxifen Citrate (pre-menopausal women) OR
    * Aromatase Inhibition Therapy (post-menopausal women)
  Interventions: Procedure: Neoadjuvant Therapy; Procedure: Therapeutic Conventional Surgery; Other: Laboratory Biomarker Analysis; Genetic: Gene Expression Analysis; Drug: Tamoxifen Citrate; Drug: Aromatase Inhibition Therapy
- Group 2 Arm 2 (RS 11-25) (Experimental): Patients with an intermediate RS(11-25) assigned to Group 2. Randomized to Arm 2, neoadjuvant chemotherapy 6-8 courses of anthracycline/taxane based regimen over 4-6 months in the absence of disease progression or unacceptable toxicity.
  Treatment:
  * Neoadjuvant therapy
  * Therapeutic conventional surgery
  * Laboratory biomarker analysis/Correlative studies
  * Gene Expression Analysis/Oncotype DX Gene Expression Profiling System
  * Systemic chemotherapy
  Interventions: Procedure: Neoadjuvant Therapy; Procedure: Therapeutic Conventional Surgery; Other: Laboratory Biomarker Analysis; Genetic: Gene Expression Analysis; Drug: Systemic Chemotherapy
- Group 3 (RS > 25) (Experimental): Patients with a high RS (> 25) assigned to Group 3, neoadjuvant chemotherapy as in Group 2 Arm 2.
  Treatment:
  * Neoadjuvant therapy
  * Therapeutic conventional surgery
  * Laboratory biomarker analysis/Correlative studies
  * Gene Expression Analysis/Oncotype DX Gene Expression Profiling System
  * Systemic chemotherapy
  Interventions: Procedure: Neoadjuvant Therapy; Procedure: Therapeutic Conventional Surgery; Other: Laboratory Biomarker Analysis; Genetic: Gene Expression Analysis; Drug: Systemic Chemotherapy

INTERVENTIONS:
Procedure: Neoadjuvant Therapy — Undergo neoadjuvant therapy
  Other Names: Induction Therapy; Neoadjuvant; Preoperative Therapy
Procedure: Therapeutic Conventional Surgery — Undergo therapeutic conventional surgery
Other: Laboratory Biomarker Analysis — Correlative studies
  Other Names: Correlative studies
Genetic: Gene Expression Analysis — Undergo Oncotype Dx gene expression profiling. The Oncotype DX gene expression profiling system will be used to calculate a "Recurrence Score" (RS).
Drug: Systemic Chemotherapy — Undergo chemotherapy
  Arms: Group 2 Arm 2 (RS 11-25); Group 3 (RS > 25)
Drug: Tamoxifen Citrate — Undergo hormonal therapy
  Other Names: Nolvadex; TAM; tamoxifen; TMX; hormonal therapy
  Arms: Group 1 (RS < 11); Group 2 Arm 1 (RS 11-25)
Drug: Aromatase Inhibition Therapy — Undergo hormonal therapy
  Other Names: Inhibition therapy, aromatase; Aromatase Inhibition; hormonal therapy
  Arms: Group 1 (RS < 11); Group 2 Arm 1 (RS 11-25)

SUMMARY:
This randomized pilot clinical trial studied whether the Oncotype DX gene expression "Recurrence Score" (RS) would be useful for helping make a decision about which type of pre-operative treatment, hormone therapy or chemotherapy would be a better for patients with hormone responsive cancers that were not suitable for breast conserving surgery. The RS is currently used to predict the risk of distant recurrence and the benefit of the addition of chemotherapy to hormonal therapy in the adjuvant setting.

DETAILED DESCRIPTION:
Assessed the feasibility of carrying out a large-scale multi-center trial in which recurrence score (RS) was used to select treatment type in the neoadjuvant setting. Whether patients with intermediate RS were willing to be randomized between hormonal and chemotherapy.

The treatment received was not experimental and considered standard treatment for the type of cancer the participants had. What was experimental included the way in which they were assigned to a type of treatment. The design of this study was used to help determine if RS can be used to predict which type of treatment women with breast cancer are most likely to benefit from.

OUTLINE: Patients are assigned to 1 of 3 groups based on RS following Oncotype Dx gene expression profiling.

* GROUP 1 (RS < 11): Patients receive neoadjuvant hormonal therapy comprising tamoxifen (pre-menopausal women) or an aromatase inhibitor (post-menopausal women) for 4-6 months in the absence of disease progression or unacceptable toxicity.
* GROUP 2 (RS 11-25): Patients are randomized to 1 of 2 treatment arms:

  * ARM 1: Patients receive neoadjuvant hormonal therapy as in group I.
  * ARM 2: Patients receive 6-8 courses of neoadjuvant chemotherapy comprising an anthracycline/taxane based regimen over 4-6 months in the absence of disease progression or unacceptable toxicity.
* GROUP 3 (RS > 25): Patients receive neoadjuvant chemotherapy as in group 2 arm 2.

All patients undergo surgery and receive hormonal therapy for at least 5 years.

After completion of study treatment, patients are followed up periodically.

ELIGIBILITY:
Inclusion Criteria:

* The treating surgeon must determine that breast conservation therapy (BCT) would be made more feasible by reducing tumor size using neoadjuvant systemic therapy
* The patient must have signed and dated an institutional review board (IRB) approved consent form that conforms to federal and institutional guidelines
* The patient must be female
* The patient must be greater than or equal to 18 years old
* The patient must have an Eastern Cooperative Oncology Group Score (ECOG) performance status of 0 or 1
* The diagnosis of invasive carcinoma of the breast must have been made by core needle biopsy
* The primary breast tumor must be >= 2 cm by physical exam or imaging
* Ipsilateral axillary lymph nodes must be evaluated by imaging (MRI or ultrasound) within 6 weeks prior to randomization; If indicated for abnormal lymph nodes, fine needle aspirate (FNA) or core biopsy must be performed.
* The tumor must have been determined to be HER2-negative as follows:

  * Fluorescent in situ hybridization (FISH)-negative (defined by ratio of HER2 to Chromosome 17 centromere (CEP17) must be < 2.2) or, if a ratio was not performed, the HER2 gene copy number must be < 4 per nucleus; or
  * Chromogenic in situ hybridization (CISH) is performed, the result must indicate a HER2 gene copy number of < 6 per nucleus; or
  * Immunohistochemistry (IHC) 0-1+; or
  * IHC 2+ and FISH-negative or CISH-negative
* The tumor must have been determined to be ER+ and/or progesterone positive (PgR+) defined as > 10% tumor staining by immunohistochemistry
* The patient must have been evaluated by a treating physician, reviewed and discussed by the multi-disciplinary breast team, and considered to be a candidate for chemotherapy

Exclusion Criteria:

* FNA alone to diagnose the primary tumor
* Excisional biopsy or lumpectomy performed prior to randomization
* Surgical axillary staging procedure or sentinel node (SN) biopsy performed prior to registration
* Tumors clinically staged as including inflammatory breast cancer
* Ipsilateral cN2b or cN3 disease (patients with cN1 or cN2a disease are eligible)
* Definitive clinical or radiologic evidence of metastatic disease (Note: chest imaging [mandatory for all patients] and other imaging [if required] must have been performed within 6 weeks prior to randomization)
* Synchronous or metachronous contralateral invasive breast cancer; (patients with synchronous and/or metachronous contralateral ductal carcinoma in situ (DCIS) or lobular carcinoma in situ (LCIS) are eligible)
* HER2 test result of IHC 3+, regardless of FISH results, if performed
* Any history of ipsilateral invasive breast cancer or ipsilateral DCIS if treated with radiation therapy (RT); (patients with synchronous or metachronous ipsilateral LCIS are eligible)
* History of non-breast malignancies, except for in situ cancers treated only by local excision and basal cell and squamous cell carcinomas of the skin, within 5 years prior to randomization
* Treatment including RT, chemotherapy, and/or targeted therapy for the currently diagnosed breast cancer prior to registration
* Cardiac disease (history of and/or active disease) that would preclude the use of chemotherapy
* Pregnancy or lactation at the time of randomization; (Note: pregnancy testing must be performed within 2 weeks prior to randomization for women of childbearing potential)
* Other non-malignant systemic disease that would preclude the patient from receiving study treatment or would prevent required follow-up
* Psychiatric or addictive disorders or other conditions that, in the opinion of the investigator, would preclude the patient from meeting the study requirements
* Use of any investigational product within 30 days prior to registration

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2011-04; Primary Completion 2015-05 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Harry D. Bear, MD, PhD, Principal Investigator — Virginia Commonwealth University
Locations (8):
- United States (7):
  - Washington Cancer Institute, Washington D.C., District of Columbia
  - Carolinas Medical Center, Charlotte, North Carolina
  - Forsyth Regional Cancer Center, Charlotte, North Carolina
  - Cone Health Cancer Center, Greensboro, North Carolina
  - Methodist Cancer Center, Houston, Texas
  - Lynchburg Hematology Oncology Clinic, Inc, Lynchburg, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
- Centre Hospitalier de l'Université de Montréal , Hôtel-Dieu Hospital, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- See also: VCU Massey Cancer Center — http://www.massey.vcu.edu/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Once a patient consented to this study and was deemed eligible the core biopsy blocks or slides were sent to obtain the Oncotype DX Breast Cancer Assay. After the Recurrence Score(RS) results were available the subject was assigned to Group 1, 2, or 3. If assigned to Group 2 they were randomized to Arm 1 or Arm 2.
Pre-assignment Details: 5/64 subjects were not assigned or randomized to an arm: delayed oncotype result, core block lost, discrepancy in a bio-marker test, and two subjects deemed not eligible. There were 5 subjects who refused assigned randomization Group 2 Arm 2. 2/5 subjects who refused Group 2 Arm 2 were treated and evaluable for response on Arm 1.
Groups:
- Group 1 (RS < 11): Patients with a RS of less than 11 were assigned to Group 1. They received neoadjuvant hormonal therapy comprised of tamoxifen (pre-menopausal women) or an aromatase inhibitor (post-menopausal women) for 4-6 months in the absence of disease progression or unacceptable toxicity.
  Treatment:
  * Neoadjuvant therapy
  * Therapeutic conventional surgery
  * Laboratory biomarker analysis/Correlative studies
  * Gene Expression Analysis/ Oncotype DX Gene Expression Profiling System
  * Hormonal therapy:
    * Tamoxifen Citrate (pre-menopausal women) OR
    * Aromatase Inhibition Therapy (post-menopausal women)
- Group 2 Arm 1 (RS 11-25): Patients with an intermediate RS (11-25) were assigned to Group 2. If randomized to Arm 1 they received neoadjuvant hormonal therapy as in Group 1.
  Treatment:
  * Neoadjuvant therapy
  * Therapeutic conventional surgery
  * Laboratory biomarker analysis/Correlative studies
  * Gene Expression Analysis/ Oncotype DX Gene Expression Profiling System
  * Hormonal therapy:
    * Tamoxifen Citrate (pre-menopausal women) OR
    * Aromatase Inhibition Therapy (post-menopausal women)
- Group 2 Arm 2 (RS 11-25): Patients with an intermediate RS (11-25) were assigned to Group 2. If randomized to Arm 2 they received 6-8 courses of neoadjuvant chemotherapy comprised of anthracycline/taxane based regimen over 4-6 months in the absence of disease progression or unacceptable toxicity.
  Treatment:
  * Neoadjuvant therapy
  * Therapeutic conventional surgery
  * Laboratory biomarker analysis/Correlative studies
  * Gene Expression Analysis/Oncotype DX Gene Expression Profiling System
  * Systemic chemotherapy
- Group 3 (RS > 25): Patients with a high RS (> 25) were assigned to Group 3. They received chemotherapy, neoadjuvant chemotherapy as in Group 2 Arm 2.
  Treatment:
  * Neoadjuvant therapy
  * Therapeutic conventional surgery
  * Laboratory biomarker analysis/Correlative studies
  * Gene Expression Analysis/Oncotype DX Gene Expression Profiling System
  * Systemic chemotherapy
Period: Recurrence Score(RS)Assigned/Randomized
Arm/Group | Group 1 (RS < 11) | Group 2 Arm 1 (RS 11-25) | Group 2 Arm 2 (RS 11-25) | Group 3 (RS > 25)
Started | 12 | 17 | 16 | 14
Assigned/Randomized to Arm | 12 | 17 | 16 | 14
Completed | 12 | 17 | 11 (2/5 subjects who refused Arm 2(chemo) were treated with Arm 1(hormonal) and evaluable for response.) | 14
Not Completed | 0 | 0 | 5 | 0
Not completed — Refused Assigned Arm | 0 | 0 | 5 | 0
Period: Treatment
Arm/Group | Group 1 (RS < 11) | Group 2 Arm 1 (RS 11-25) | Group 2 Arm 2 (RS 11-25) | Group 3 (RS > 25)
Started | 12 | 19 (2/5 subjects who refused Arm 2(chemo) were treated with Arm 1(hormonal) and evaluable for response.) | 11 | 14
Completed | 10 | 14 | 10 | 13
Not Completed | 2 | 5 | 1 | 1
Not completed — Adverse Event | 0 | 0 | 1 | 1
Not completed — Withdrawal by Subject | 2 | 4 | 0 | 0
Not completed — Disease Progression, relapse | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Group 1 (RS < 11): Patients with a Recurrence Score (RS) of less than 11 were assigned to Group 1. They received neoadjuvant hormonal therapy comprised of tamoxifen (pre-menopausal women) or an aromatase inhibitor (post-menopausal women) for 4-6 months in the absence of disease progression or unacceptable toxicity.
  Treatment:
  * Neoadjuvant therapy
  * Therapeutic conventional surgery
  * Laboratory biomarker analysis/Correlative studies
  * Gene Expression Analysis/ Oncotype DX Gene Expression Profiling System
  * Hormonal therapy:
    * Tamoxifen Citrate (pre-menopausal women) OR
    * Aromatase Inhibition Therapy (post-menopausal women)
- Total: Total of all reporting groups
Arm/Group | Group 1 (RS < 11) | Group 2 Arm 1 (RS 11-25) | Group 2 Arm 2 (RS 11-25) | Group 3 (RS > 25) | Total
Number analyzed (Participants) | 12 | 17 | 16 | 14 | 59
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 5 | 8 | 13 | 10 | 36
  >=65 years | 7 | 9 | 3 | 4 | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.3125 (5.931426) | 63.64706 (11.5539) | 55.3125 (12.2556) | 60.64286 (7.312867) | 61.25423729 (10.52188724)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 17 | 16 | 14 | 59
  Male | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1 | 0 | 2
  Not Hispanic or Latino | 11 | 16 | 15 | 14 | 56
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 5 | 0 | 4 | 2 | 11
  White | 7 | 17 | 12 | 12 | 48
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Canada | 1 | 4 | 2 | 4 | 11
  United States | 11 | 13 | 14 | 10 | 48

OUTCOME MEASURES:

1. Primary Outcome: The Proportion of Patients With RS 11-25 Who Refused the Assigned Treatment
Description: The primary purpose of this trial is to determine the feasibility of carrying out a large multi-center trial with a similar design. Feasibility, in terms of less than 1/3 of patients with intermediate (11-25) Recurrence Score (RS) who refused the assigned treatment (Group 2) or refused randomization between hormonal (Arm 1) or chemotherapy (Arm 2). The confidence interval will be 95%. The proportion (and 95% confidence interval) of patients with RS 11-25 who refuse the assigned treatment will be calculated.
Time Frame: Up to 2 years
Population: Patients with an intermediate RS(11-25) assigned to Group 2, Arm 1, and Arm 2 were combined in the analysis.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Groups:
- Group 2 (RS 11-25): Patients with an intermediate RS (11-25) were assigned to Group 2. The subject was then randomized to treatment Arm 1, neoadjuvant hormonal therapy, or treatment Arm 2, neoadjuvant chemotherapy.
Arm/Group | Group 2 (RS 11-25)
Number analyzed (Participants) | 33
proportion of participants | 0.15 [0.051 to 0.319]

ADVERSE EVENTS:
Description: Adverse events (AEs) that are a result of standard diagnosis and treatment are not being collected and should not be reported.
Arm/Group | Group 1 (RS < 11) | Group 2 Arm 1 (RS 11-25) | Group 2 Arm 2 (RS 11-25) | Group 3 (RS > 25)
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes